CLINICAL TRIAL: NCT01886365
Title: Perioperative Glycemic Control With a Computerized Algorithm vs. Conventional Glycemic Control in Cardio-surgical Patients Undergoing Cardiopulmonary Bypass With Blood Cardioplegia
Brief Title: Computerized Tight Glycemic Control in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Daniel Reuter, Professor of anesthesiology, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV3388
Record Dates: First submitted 2013-06-12; First posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Hyperglycemia
Keywords: Computer based glycemic control, insulin, blood glucose
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): With start of the cardiopulmonary bypass, computerized algorithmic application of insulin was performed with a dedicated computerized syringe pump system (Space GlucoseControl System, B. Braun, Germany). The targeted corridor for blood glucose was determined with 80 - 150 mg/dl. During surgery, blood glucose was measured every 30 min, and on the ICU every 2 hours. TGC management was continued until ICU discharge.
  Interventions: Device: Space GlucoseControl System, B. Braun, Melsungen, Germany
- Group B (Active Comparator): Corresponding computerized algorithmic application of insulin management was used as for group A. However, only the interval of blood glucose measurement during surgery was adjusted to 15 minutes.
  Interventions: Device: Space GlucoseControl System, B. Braun, Melsungen, Germany
- Group C (Other): With start of the cardiopulmonary bypass conventional therapy with a fixed insulin dosing scheme was initiated. If blood glucose was > 150 mg/dl, manual insulin therapy was started following a fixed insulin dosing scheme. Measurements of blood glucose were performed during surgery every 30 minutes, and on the ICU every 2 hours until discharge (Routine Care).
  Interventions: Other: Conventional therapy with a fixed insulin dosing scheme

INTERVENTIONS:
Device: Space GlucoseControl System, B. Braun, Melsungen, Germany — Computerized algorithmic application of insulin
  Arms: Group A; Group B
Other: Conventional therapy with a fixed insulin dosing scheme — Routine care
  Arms: Group C

SUMMARY:
The debate about tight glycemic control (TGC) in the operating room and on the intensive care unit is ongoing, especially in cardio-surgical patients treated with blood cardioplegia, due to high blood glucose levels during operations and subsequent high rates of sternal wound infections. We showed in a feasibility study that early computer based insulin therapy starting in the operating room is a safe therapy that allows to better warrant normoglycemia in patients undergoing major cardiac surgery with the use of blood cardioplegia.

DETAILED DESCRIPTION:
Patients are enrolled and randomized into 3 groups. Start of therapy is determined as the beginning of cardiopulmonary bypass. Group A: Therapy with computer-based algorithm and measurement of blood glucose every 30 min. Group B: Measurement of blood glucose every 15 min using the identical computer-based algorithm. Group C: Conventional therapy using a fixed insulin dosing scheme. End of therapy is defined as discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 scheduled for elective cardiac surgery with the use of cardiopulmonary bypass and blood cardioplegia

Exclusion Criteria:

* under 18 years of age, or if patients had a premedical history of steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time within a blood glucose corridor of 80 - 150 mg/dl | From start of cardiopulmonary bypass during surgery until discharge from ICU, which is approximately after 48 -72 hrs.
  The primary endpoint was defined as the time within a given blood glucose corridor from 80 - 150 mg/dl during therapy

SECONDARY OUTCOMES:
Hypoglycemic events | From beginning of cardiopulmonary bypass during surgery until discharge from the ICU, which is approximately after 48-72 hrs.
  Secondary endpoints were the number of hypoglycemic events defined as blood glucose levels under 80 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Reuter, Professor, Principal Investigator — University Medical Center Hamburg-Eppendorf, Germany
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Punke MA, Goepfert MS, Kluge S, Reichenspurner H, Goetz AE, Reuter DA. Perioperative glycemic control with a computerized algorithm versus conventional glycemic control in cardiac surgical patients undergoing cardiopulmonary bypass with blood cardioplegia. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1273-7. doi: 10.1053/j.jvca.2014.04.017. PMID 25281044